CLINICAL TRIAL: NCT03114800
Title: Monitoring Movement for Pressure Ulcer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Pearlman (Other)
Responsible Party: Sponsor-Investigator, Jonathan Pearlman, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PRO16120412
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- E-Scale (Experimental): Weight monitoring
  Interventions: Device: E-Scale

INTERVENTIONS:
Device: E-Scale — The E-Scale is comprised of a series of weight monitoring 'pods' and a set of software modules that facilitate data transfer and analysis.
  Other Names: Embedded Scale

SUMMARY:
The goal of this work is to develop and test an automated movement detection monitoring tool that could lead to reduced burden on clinicians and in-turn reduce pressure ulcer incidence rates. Ten healthy participants will perform video-recorded bed movements while weight distribution and interface pressures at bony prominences on the pelvis are recorded.

DETAILED DESCRIPTION:
The incidence rate and subsequent costs of preventable pressure ulcers is astounding. Although pressure ulcer risk assessment tools and prevention approaches have been a topic of research and for many years, the incidence rate has remained relatively consistent. One reason that progress has not been made to lower the incidence rate is that there is no objective monitoring tool to determine how much a person is moving or is being moved in their bed. Current practices are time-intensive and have not yet leveraged intelligent monitoring technology that could reduce clinical burden and increase accuracy of the risk assessment and efficacy of prevention protocols. The goal of this work is to develop and test an automated movement detection monitoring tool that could lead to reduced burden on clinicians and in-turn reduce pressure ulcer incidence rates. This monitoring tool will be an extension of our intelligent bed sensor we developed named the Embedded Scale, or E-Scale. The E-Scale currently has software modules that detect bed exit, individual weight, and multi-person weight. The project described here would develop a movement module for the E- Scale to monitor people's movements in bed in an attempt to eventually reduce incidence of pressure ulcers in clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older

Exclusion Criteria:

* Not able to independently get onto a bed and reposition themselves
* Skin lesions in the area where sensors will be placed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Weight change | 1 hour
  Weight change at each load cell

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Pearlman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Bakery Square, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will be used to develop a proprietary algorithm